CLINICAL TRIAL: NCT06311019
Title: The Effects of Continuous Glucose Monitoring and Connected Insulin Pens on Glycemic Control in Patients With Type 2 Diabetes Treated With Multiple Daily Insulin Injections.
Brief Title: The Effects of CGM and Connected Pen in T2DM Treated With Multiple Daily Insulin Injections
Acronym: Dia2tech
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Klavs Würgler Hansen (Other)
Collaborators: Steno Diabetes Center Aarhus, Denmark (Unknown)
Responsible Party: Sponsor-Investigator, Klavs Würgler Hansen, Professor, Central Jutland Regional Hospital
Organization: Central Jutland Regional Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 791572
Record Dates: First submitted 2024-02-06; First posted 2024-03-15 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Type 2 Diabetes Treated With Insulin
Keywords: Type 2 diabetes mellitus; Insulin; Continuous glucose monitoring; Connected Pen
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Standard care) (No Intervention): In this arm the patients continue to measure blood glucose with fingerprick and use standard insulin pens
- 2 (CGM and connected pen) (Active Comparator): In this arm the patients switch from glucose measurement with fingerprick to continuous glucose monitoring and they switch from standard insulin pen for bolusinsulin to connected pen for bolusinsulin
  Interventions: Device: Continuous glucose monitoring and use of connected insulinpen for bolus insulin

INTERVENTIONS:
Device: Continuous glucose monitoring and use of connected insulinpen for bolus insulin — Continuous glucose monitoring (Abbott Freestyle Libre 2) and use of connected insulinpen (Novopen 6) for bolus insulin
  Arms: 2 (CGM and connected pen)

SUMMARY:
The aim of the study is to evaluate the effect of a combination of 12 months treatment with CGM (Freestyle Libre 2) with hypo and hyper alert in combination with a smart pen for bolus insulin (NOVOpen6) on HbA1c and time in range (TIR) in T2DM patients with baseline HbA1c >53 mmol/mol (7. 0%, eAG 8,6 mmol/l) as compared with standard care.

DETAILED DESCRIPTION:
This study is a 12 months open-label randomized controlled trial.

Subjects with basal/bolus insulin treated T2DM and HbA1c >53 mmol/mol are randomized to:

A (control): standard care with disposable insulin pens and fingerprick glucose measurement or B (intervention): Novopen6 for bolus insulin and glucose measurement with Freestyle Libre 2.

Due to the nature of the treatments it is not possible to perform a blinded study.

Randomization in ratio 1:1 will be formed electronically in a REDCap database.

The investigators estimate that the mean HbA1c at baseline is 60 mmol/mol. Given a standard deviation of the difference of approximately 8.1 mmol/mol (based on in house data from 114 patients with T2DM and insulin), the investigators calculate that 47 patients are needed in each arm to detect a minimal relevant difference of 5 mmol/mol with a type I error of 5% and a type II error 15%. Allowing for 10 % dropouts, the investigators aim to recruit 52 patients in each arm. If an interim analysis 3 months after randomizing 40 patients suggest a higher drop-out rate, the study size will be increased accordingly to a drop-out rate of max. 20 % (56 in each arm).

Study plan

Pre-screening of eligible patients was performed by assessing data from the healthcare administrative electronic software platform Business Intelligence (BI) of the Central Denmark Region. In this portal, data on medication, lab results, time period for contact to outpatient clinic for persons followed in secondary healthcare are automatically registered by data capture. Data can be retrieved from the BI portal via access to an encrypted version of the civil registration numbers allocated to all Danish citizens. The investigators collected data on prescribed pharmacological treatment for all persons with Type 2 diabetes who have had a minimum of one contact to the study centers.

The electronic patient records for potential study candidates were reviewed for in- and exclusion criteria. Patients still considered study candidates after pre-screening were contacted by e-mail and invited to a meeting.

Visit 1 (- 4 weeks): Inclusion and exclusion criteria are reviewed. Orally information of the study plan provided with reflection-time up to 24 hours. Planning fasting blood sample, blinded CGM (Freestyle Libre Pro) is applied, medication reviewed. Questionnaires answered.

Visit 2 (-2 weeks): Fasting blood samples, Libre Pro removed and uploaded.

Visit 3 (0 months): Randomization if inclusion criteria are full-filled and no exclusion criteria. Otherwise considered a screening failure. Randomization to either:

A (control): continues treatment with usual insulin pens and self measurements of blood glucose.

B (intervention): changes to NovoPen 6 for bolus insulin and CGM (Abbott Freestyle Libre 2). Patients randomized to intervention will participate in a structured education programme about the clinical use of Libre 2 and Novopen 6. This also includes assistance to upload LibreLink app. on the mobile phone, to upload Novopen 6 data and to establish a Libre View account. The patients fill in the diabetes health related questionnaires.

Visit 4 Intervention group only (1 month): Telephone call (by study nurse) or optional personal meeting as necessary. Technical support only as needed for the upload of Freestyle Libre 2 and Novopen6 to LibreView.

Visit 5 (11½ months): Blinded Freestyle Libre Pro is applied to all subjects (arm A and B).

Visit 6 (12 months): Blood sample for HbA1c. Discontinuation and upload of Freestyle Libre Pro IQ (Libre view) and blood glucose-meter (Glooko)) for the last 14 days for both the control and intervention arm. In addition upload of Libre 2 and Novopen6 data (Libre view) for the last 4 weeks is performed for the intervention arm. Fill in of diabetes health related questionnaires and use of the memory function of Novopen 6

In-between study visits patients follow standard care in terms of number of visits (physical or telemedicine), type of health care provider (nurse or doctor), measurement of HbA1c and other clinical activities at the health care providers discretion, to enhance extern validity.

The glucose data is evaluated by the usual health care providers together with the patient in order to optimize insulin therapy, including an increase in the number of meals with bolus insulin if necessary.

According to the study design all patients are treated with bolus insulin for at least one meal. Bolus insulin should be insulin aspart. If patients are treated with insulin aspart manufactured by other companies than Novo Nordisk, the patients are asked to change to the biosimilar product from Novo. This strategy ensures that all patients can undergo randomization, since only Novo products fits into the Novopen6. Fast acting insulin is provided to all the patients in the study period free of charge. Patients randomized to the intervention group B receives Novopen6 free of charge.

Patients are included irrespective of the brand of basal insulin. Any other glucose lowering drug (oral or injection) can be added or discontinued during the study at the investigators discretion.

ELIGIBILITY:
Inclusion Criteria:

1. - Type 2 DM.
2. - HbA1c > 53 mmol/l (7.0 %, estimated average glucose (eAG) 8.6 mmol/l).
3. - Contact to diabetes clinic for ≥ 6 months.
4. - Insulin treatment ≥ 12 months.
5. - Basal insulin and bolus insulin at least for one meal every day.
6. - Bolus insulin is insulin aspart.
7. - Stable insulin treatment (change 10 % or less) and no introduction of other antihyperglycemic agents (oral or GLP1 analogue) for at least 2 months before randomization.
8. - Considered to be technically and intellectually capable of using isCGM and smart pen.
9. - Can communicate in Danish.
10. - Informed consent including acceptance to share glucose data from the Libreview platforms.
11. - The patient has a smart phone suitable for Libre and NOVOpen6 data registration.

Exclusion Criteria:

1. - Individual goal for HbA1c is reached (even if > 53 mmol/mol), i.e. relaxed treatment goals as relevant for fragile patients with severe diabetic complications or comorbidities.
2. - Fasting C-peptide < 370 pmol/l.
3. - Actual treatment with CGM or previous use of CGM for more than four weeks or < 6 months before recruitment. No actual or previous use of connected pen.
4. - One or more severe hypoglycemic episode (assistance of third party) within the previous 12 months.
5. - Considered unable to participate due to frequent cancellation of appointments.
6. - Ongoing steroid treatment or expected intermittent treatment of more than 14 days' duration.
7. - Pregnant or planning pregnancy.
8. - Participating in other trials.
9. - Clinical conditions interfering with interpretation of HbA1c (phlebectomy, bleeding or haemolytic disorders, erythropoietin treatment, known haemoglobin variants, etc.) or continuous intake of high dose of vitamin C (> 1000 mg), salicylic acid (650 mg daily), Salazopyrin or Dapsone.
10. - Allergic reaction to the adhesive used in the isCGM.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Haemoglobin A1c | Baseline and follow-up after 12 months
  Change between groups in Haemoglobin A1c (mmol/mol) from baseline to follow-up
  A prespecified exploratory analysis is planned for:
  male vs. female age < 65 year vs. age ≥ 65 year baseline HbA1c < 58 mmol/l vs baseline HbA1c ≥58 mmol/l Bolus insulin for 1 or 2 meals at baseline vs. bolus insulin for > 2 meals Number of average views by Libre 2 for the last month < 10 vs. per day vs. ≥10 scannings.
  A per-protocol analysis will be performed for patients in the intervention arm with available glucose values for more than 70 % of the time during the last 30 days.

SECONDARY OUTCOMES:
Change Time in range | Baseline and follow-up after 12 months
  Change in the fraction (%) of glucose values in the range 3.9 to 10.0 mmol/l, measured by Libre Pro IQ for 14 days.
  A prespecified exploratory analysis is planned for:
  male vs. female age < 65 year vs. age ≥ 65 year baseline HbA1c < 58 mmol/l vs baseline HbA1c ≥58 mmol/l Bolus insulin for 1 or 2 meals at baseline vs. bolus insulin for > 2 meals Number of average views by Libre 2 for the last month < 10 vs. per day vs. ≥10 scannings.
  A per-protocol analysis will be performed for patients in the intervention arm with available glucose values for more than 70 % of the time during the last 30 days.
Change in Time above range | Baseline and follow-up after 12 months
  Change in The fraction (%) of glucose values in the range > 10.0 mmol/l, measured by Libre Pro IQ for 14 days.
  A prespecified exploratory analysis is planned for:
  male vs. female age < 65 year vs. age ≥ 65 year baseline HbA1c < 58 mmol/l vs baseline HbA1c ≥58 mmol/l Bolus insulin for 1 or 2 meals at baseline vs. bolus insulin for > 2 meals Number of average views by Libre 2 for the last month < 10 vs. per day vs. ≥10 scannings.
  A per-protocol analysis will be performed for patients in the intervention arm with available glucose values for more than 70 % of the time during the last 30 days.
Change in Time below range | Baseline and follow-up after 12 months
  Change in the fraction (%) of glucose values < 3.9 mmol/l, measured by Libre Pro IQ for 14 days.
  A prespecified exploratory analysis is planned for:
  male vs. female age < 65 year vs. age ≥ 65 year baseline HbA1c < 58 mmol/l vs baseline HbA1c ≥58 mmol/l Bolus insulin for 1 or 2 meals at baseline vs. bolus insulin for > 2 meals Number of average views by Libre 2 for the last month < 10 vs. per day vs. ≥10 scannings.
  A per-protocol analysis will be performed for patients in the intervention arm with available glucose values for more than 70 % of the time during the last 30 days.
Mean glucose | Baseline and follow-up after 12 months
  The mean of all glucose values for 14 days measured by Libre Pro IQ.
  A prespecified exploratory analysis is planned for:
  male vs. female age < 65 year vs. age ≥ 65 year baseline HbA1c < 58 mmol/l vs baseline HbA1c ≥58 mmol/l Bolus insulin for 1 or 2 meals at baseline vs. bolus insulin for > 2 meals Number of average views by Libre 2 for the last month < 10 vs. per day vs. ≥10 scannings.
  A per-protocol analysis will be performed for patients in the intervention arm with available glucose values for more than 70 % of the time during the last 30 days.
Standard deviation | Baseline and follow-up after 12 months
  The standard deviation of glucose values for 14 days, measured by Libre Pro IQ.
  A prespecified exploratory analysis is planned for:
  male vs. female age < 65 year vs. age ≥ 65 year baseline HbA1c < 58 mmol/l vs baseline HbA1c ≥58 mmol/l Bolus insulin for 1 or 2 meals at baseline vs. bolus insulin for > 2 meals Number of average views by Libre 2 for the last month < 10 vs. per day vs. ≥10 scannings.
  A per-protocol analysis will be performed for patients in the intervention arm with available glucose values for more than 70 % of the time during the last 30 days.
Change in CV | Baseline and follow-up after 12 months
  Change in the coefficient of variation (%) for glucose values for 14 days, measured by Libre Pro IQ for 14 days.
  A prespecified exploratory analysis is planned for:
  male vs. female age < 65 year vs. age ≥ 65 year baseline HbA1c < 58 mmol/l vs baseline HbA1c ≥58 mmol/l Bolus insulin for 1 or 2 meals at baseline vs. bolus insulin for > 2 meals Number of average views by Libre 2 for the last month < 10 vs. per day vs. ≥10 scannings.
  A per-protocol analysis will be performed for patients in the intervention arm with available glucose values for more than 70 % of the time during the last 30 days.
Change in Time with rapid glucose change | Baseline and follow-up after 12 months
  Change in the time fraction (%) with glucose rate of change > 1.5 mmol/l/15 min, measured by Libre Pro. A prespecified exploratory analysis is planned for:
  male vs. female age < 65 year vs. age ≥ 65 year baseline HbA1c < 58 mmol/l vs baseline HbA1c ≥58 mmol/l Bolus insulin for 1 or 2 meals at baseline vs. bolus insulin for > 2 meals Number of average views by Libre 2 for the last month < 10 vs. per day vs. ≥10 scannings.
  A per-protocol analysis will be performed for patients in the intervention arm with available glucose values for more than 70 % of the time during the last 30 days.
  IQ for 14 days.
Change in ARRC | Baseline and follow-up after 12 months
  Change in Mean of average absolute change of glucose rate (ml/mol/15 min), measured by Libre Pro IQ for 14 days. A prespecified exploratory analysis is planned for:
  male vs. female age < 65 year vs. age ≥ 65 year baseline HbA1c < 58 mmol/l vs baseline HbA1c ≥58 mmol/l Bolus insulin for 1 or 2 meals at baseline vs. bolus insulin for > 2 meals Number of average views by Libre 2 for the last month < 10 vs. per day vs. ≥10 scannings.
  A per-protocol analysis will be performed for patients in the intervention arm with available glucose values for more than 70 % of the time during the last 30 days.
Fraction of patients with increased number of bolus insulin per day | Baseline and follow-up after 12 months
  The fraction of patients increasing from one or two meals with bolus insulin to two or three meals with bolus insulin.

OTHER OUTCOMES:
Fingerprick glucose measurement | Baseline and follow-up after 12 months
  Number of fingerprick glucose measurements for the last 14 days.(fromGlooko download) of BG meters)
Glucose views on mobile phone | Follow-up at 12 months
  Numbers of glucose views in the last 14 days in the intervention group (from LibreView).
Use of Novopen 6 memory function | Follow-up at 12 months
  Self reported numbers of inspections of the insulindose/time on the Novopen 6 cap display for the last 14 days in the intervention group.
WHO-5 | Baseline and follow-up at 12 months
  Questionnaire
Diabetes Distress Scale | Baseline and follow-up at 12 months
  Questionnaire
Revised short form of hypoglycaemia Fear Survey | Baseline and follow-up at 12 months
  Questionnaire
eHealth literacy questionnaire (eHLQ), | Baseline and follow-up at 12 months
  Questionnaire
The Glucose Monitoring Satisfaction Questionnaire | Baseline and follow-up at 12 months
  Questionnaire
Diabetes Treatment Satisfaction Questionnaire (DTSQ) | Baseline and follow-up at 12 months
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Klavs W Hansen, Study Director — Medical Diagnostic Center, Silkeborg Regional Hospital
Locations (5):
- Denmark (5):
  - Steno Diabetes Center Aarhus, Aarhus
  - Gødstrup Regional Hospital, Herning
  - Horsens Regional Hospital, Horsens
  - Randers Regional Hospital, Randers
  - Regional Hospital Silkeborg, Central Jutland Hospital, Silkeborg

IPD SHARING:
Plan to Share IPD: Yes
Data planned to make available: All primary and secondary outcome values
Supporting Information: Study Protocol, CSR
Time Frame: 2026
Access Criteria: on reasonable request